CLINICAL TRIAL: NCT06239116
Title: A Study of RM-718 Weekly Formulation in Healthy Subjects With Obesity and in Patients With Obesity Due to MC4R Impairment
Brief Title: A Study of RM-718 in Healthy Subjects and Patients With MC4R Pathway Impairment
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RM-718-001
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Hypothalamic Obesity; Prader-Willi Syndrome; PWS
Keywords: melanocortin 4 receptor (MC4R); MC4R agonism; obesity
MeSH Terms: conditions — Sexual Infantilism; Prader-Willi Syndrome; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study Parts A and B are blinded. Study Parts C and D are open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (17):
- RM-718 (Cohort A1) (Experimental): Single dose of RM-718 (4) or placebo (2)
  Interventions: Drug: Part A: RM-718 or placebo (matched to specific RM-718 dose cohort)
- RM-718 (Cohort A2) (Experimental): Single dose of RM-718 (4) or placebo (2)
  Interventions: Drug: Part A: RM-718 or placebo (matched to specific RM-718 dose cohort)
- RM-718 (Cohort A3) (Experimental): Single dose of RM-718 (4) or placebo (2)
  Interventions: Drug: Part A: RM-718 or placebo (matched to specific RM-718 dose cohort)
- RM-718 (Cohort A4) (Experimental): Single dose of RM-718 (4) or placebo (2)
  Interventions: Drug: Part A: RM-718 or placebo (matched to specific RM-718 dose cohort)
- RM-718 (Cohort A5) (Experimental): Single dose of RM-718 (4) or placebo (2)
  Interventions: Drug: Part A: RM-718 or placebo (matched to specific RM-718 dose cohort)
- RM-718 (Cohort A6) (Experimental): Single dose of RM-718 (4) or placebo (2)
  Interventions: Drug: Part A: RM-718 or placebo (matched to specific RM-718 dose cohort)
- RM-718 (Cohort A7) (Experimental): Single dose of RM-718 (4) or placebo (2)
  Interventions: Drug: Part A: RM-718 or placebo (matched to specific RM-718 dose cohort)
- RM-718 (Cohort A8) (Experimental): Single dose of RM-718 (4) or placebo (2)
  Interventions: Drug: Part A: RM-718 or placebo (matched to specific RM-718 dose cohort)
- RM-718 (Cohort A9) (Experimental): Single dose of RM-718 (4) or placebo (2)
  Interventions: Drug: Part A: RM-718 or placebo (matched to specific RM-718 dose cohort)
- RM-718 (Cohort B1) (Experimental): Multiple ascending doses of RM-718 (4) or placebo (2)
  Interventions: Drug: Part B: RM-718 or placebo (matched to specific RM-718 dose cohort)
- RM-718 (Cohort B2) (Experimental): Multiple ascending doses of RM-718 (4) or placebo (2)
  Interventions: Drug: Part B: RM-718 or placebo (matched to specific RM-718 dose cohort)
- RM-718 (Cohort B3) (Experimental): Multiple ascending doses of RM-718 (4) or placebo (2)
  Interventions: Drug: Part B: RM-718 or placebo (matched to specific RM-718 dose cohort)
- RM-718 (Cohort B4) (Experimental): Multiple ascending doses of RM-718 (4) or placebo (2)
  Interventions: Drug: Part B: RM-718 or placebo (matched to specific RM-718 dose cohort)
- RM-718 (Cohort B5) (Experimental): Multiple ascending doses of RM-718 (4) or placebo (2)
  Interventions: Drug: Part B: RM-718 or placebo (matched to specific RM-718 dose cohort)
- RM-718 (Cohort B6) (Experimental): Multiple ascending doses of RM-718 (4) or placebo (2)
  Interventions: Drug: Part B: RM-718 or placebo (matched to specific RM-718 dose cohort)
- RM-718 (Cohort C1) (Experimental): Multiple ascending doses of RM-718 (30)
  Interventions: Drug: Part C: RM-718
- RM-718 (Cohort D1) (Experimental): Multiple ascending doses of RM-718 (up to 30)
  Interventions: Drug: Part D: RM-718

INTERVENTIONS:
Drug: Part A: RM-718 or placebo (matched to specific RM-718 dose cohort) — Single ascending dose of RM-718 or placebo (matched to specific RM-718 Part A dose cohort)
  Arms: RM-718 (Cohort A1); RM-718 (Cohort A2); RM-718 (Cohort A3); RM-718 (Cohort A4); RM-718 (Cohort A5); RM-718 (Cohort A6); RM-718 (Cohort A7); RM-718 (Cohort A8); RM-718 (Cohort A9)
Drug: Part B: RM-718 or placebo (matched to specific RM-718 dose cohort) — Multiple ascending doses of RM-718 or placebo (matched to specific RM-718 Part B dose cohorts)
  Arms: RM-718 (Cohort B1); RM-718 (Cohort B2); RM-718 (Cohort B3); RM-718 (Cohort B4); RM-718 (Cohort B5); RM-718 (Cohort B6)
Drug: Part C: RM-718 — Multiple ascending doses of RM-718
  Arms: RM-718 (Cohort C1)
Drug: Part D: RM-718 — Multiple ascending doses of RM-718
  Arms: RM-718 (Cohort D1)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and PK of RM-718 in healthy subjects with obesity and in patients with MC4R Pathway Impairment

DETAILED DESCRIPTION:
This is a first-in-human and first-in-patient, 4-part study that includes the evaluation of safety, tolerability, and PK of: single ascending doses (SAD) of RM-718 weekly (RM-718) in healthy subjects 18 to 55 years of age with obesity (Part A), multiple ascending doses (MAD) of RM-718 in healthy subjects 18 to 55 years of age with obesity (Part B), MAD of RM-718 in patients 12 to 65 years of age with HO (Part C), and MAD of RM-718 in patients with PWS (Part D). Cohorts in Parts A and B are double-blind, placebo-controlled, and randomized 2:1 (4 subjects receive RM-718, 2 subjects receive placebo). Part C evaluates open-label dose escalation in patients 12 to 65 years of age with HO. Part D evaluates open-label dose escalation in patients 12 to 65 years of age. Study participants will receive: 1 weekly dose of either RM-718 or placebo in Part A, 4 weekly doses of either RM-718 or placebo in Part B,16 weekly doses of open-label RM-718 in Part C, and 26 weekly doses of RM-718 in Part D. Study drug (RM-718 or placebo) doses are administered weekly via subcutaneous injection.

ELIGIBILITY:
Key Inclusion Criteria:

Parts A and B:

* Male and female subjects in good health aged 18-55 years of age at Screening.
* Body mass index (BMI) ≥30 kg/m2.
* Subjects who are medically healthy with normal or clinically insignificant screening results.
* Subjects must use a highly effective form of contraception and follow the study contraception requirements.
* Ability to communicate well with the Investigator, understand and comply with the requirements of the trial, and understand English and sign the written informed consent.

Part C:

* Male and female patients with HO, aged 12-65 years of age at Screening.
* Patient has documented evidence of acquired HO defined as:

  * Diagnosis of craniopharyngioma or other brain lesion affecting the hypothalamic region and has undergone surgery, or chemotherapy, or radiation therapy involving the hypothalamus at least 6 months before Screening, OR
  * Documented injury to the hypothalamus at least 6 months before Screening for which surgery/radiation is not indicated.
* Weight gain associated with the hypothalamic injury either before or following therapy (surgery and/or following chemotherapy or radiotherapy), and a BMI of ≥30 kg/m2 for patients ≥18 years of age or BMI ≥95th percentile for age and sex for patients 12 to <18 years of age.
* Patients must use a highly effective form of contraception and follow the study contraception requirements.
* Ability to communicate with the Investigator, understand and comply with the requirements of the trial, and understand and sign the written informed consent and assent (for patients aged <18 years), and informed consent for a parent or guardian of any patient <18.

Part D:

* Confirmed diagnosis of PWS as determined by the Investigator at the time of Screening.
* Age ≥12 to 65, inclusive, at the time of signing Informed Consent and/or Assent.
* BMI ≥30 kg/m2 for patients ≥18 years of age or BMI ≥95th Percentile for age and sex for patients <18 years of age based on the US CDC criteria.
* Able to meet contraception requirements.

Key Exclusion Criteria:

Parts A and B

* Any clinically significant abnormalities on screening laboratories or physical examination as determined by the Investigator.
* Active or history of any significant medical condition such as and including renal, hepatic, pulmonary, gastrointestinal, cardiovascular, genitourinary, endocrine, immunologic, metabolic, neurologic or hematological disease.
* Obesity due to genetic, syndromic, or endocrine etiologies.
* History of renal transplant, end stage renal disease.
* Diagnosis of severe psychiatric disorders.
* Current, clinically significant pulmonary, cardiac, metabolic, or oncologic disease considered severe enough to interfere with the trial and/or confound the results.
* Cigarette smoking or dependence on caffeine, alcohol or drugs; unable or unwilling to abstain completely from caffeine, alcohol and related substances for 24 hours prior to and after study visits.
* History of recent surgery (within 60 days of Screening).
* Participation in any clinical trial with an investigational drug/device within 3 months or 5 half-lives, whichever is longer, prior to the first trial dose.
* Pregnant and/or breastfeeding or desiring to become pregnant during this trial.

Part C

* Diagnosis of Prader-Willi syndrome (PWS) or Rapid-onset obesity with hypoventilation, hypothalamic, autonomic dysregulation, neuroendocrine tumor syndrome (ROHHADNET).
* Weight loss >2% in the previous 3 months for patients aged ≥18 years or >2% reduction in BMI for patients aged 12 to <18 years and/or anti-obesity medications for the treatment of obesity.
* Bariatric surgery or procedure within the last 2 years.
* Diagnosis of severe psychiatric disorders; any suicidal ideation, attempt or behavior.
* Current, clinically significant pulmonary, cardiac, metabolic, or oncologic disease considered severe enough to interfere with the trial and/or confound the results.
* History of renal transplant, end stage renal disease.
* Participation in any clinical trial with an investigational drug/device within 3 months or 5 half-lives, whichever is longer, prior to the first trial dose, or previous participation in a trial with setmelanotide.
* Pregnant and/or breastfeeding or desiring to become pregnant during this trial.
* Obesity attributable to other genetic or syndromic conditions (eg, PPL [pro-opiomelanocortin (POMC), proprotein convertase subtilisin/kexin type 1 (PCSK1), leptin receptor (LEPR), collectively], Bardet-Biedl syndrome [BBS]) prior to the hypothalamic injury.

Part D

* Weight loss >2% in the previous 3 months for patients aged ≥18 years or >2% reduction in BMI for patients aged 12 to <18 years or therapies for the treatment of obesity or hyperphagia.
* Metabolic and bariatric surgery (MBS) or procedure within last 6 months.
* Diagnosis of severe psychiatric disorders; any suicidal ideation, attempt or behavior.
* Current, clinically significant pulmonary, cardiac, metabolic, or oncologic disease considered severe enough to interfere with the trial and/or confound the results.
* Pregnant and/or breastfeeding or desiring to become pregnant during this trial.

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Parts A, B, C, D: Safety and Tolerability Assessed by Number of Study Participants with Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From Day 1 through the Safety-Follow-up call (up to Day 43 for all Part A cohorts, up to Day 70 for all Part B cohorts, up to Day 140 for Part C cohort, up to Day 210 for Part D cohort)

SECONDARY OUTCOMES:
AUCtau measurement of RM-718 | up to 168 hours post-dose on Day 1 (Parts A, B and C) and 168 hours post-dose on Day 22 (Parts B and C).
  Area under the concentration versus time curve during a dosing interval
Cmax measurement of RM-718 | up to 168 hours post-dose on Day 1 (Parts A, B and C) and 168 hours post-dose on Day 22 (Parts B and C).
  Maximum concentration measurement of RM-718 in plasma
Cmin measurement of RM-718 | up to 168 hours post-dose on Day 1 (Parts A, B and C) and 168 hours post-dose on Day 22 (Parts B and C).
  Minimum plasma concentration of RM-718 reached during dosing interval
Tmax measurement of RM-718 | up to 168 hours post-dose on Day 1 (Parts A, B and C) and 168 hours post-dose on Day 22 (Parts B and C).
  Time it takes for RM-718 to reach the maximum concentration (Cmax)
Tmin measurement of RM-718 | up to 168 hours post-dose on Day 1 (Parts A, B and C) and 168 hours post-dose on Day 22 (Parts B and C).
  Time at which the lowest concentration value of RM-718 is observed
Ctrough measurement of RM-718 | up to 168 hours post-dose on Day 1 (Parts A, B and C) and 168 hours post-dose on Day 22 (Parts B and C).
  Observed pre-dose plasma concentration of RM-718
Cavg measurement of RM-718 | up to 168 hours post-dose on Day 1 (Parts A, B and C) and 168 hours post-dose on Day 22 (Parts B and C).
  Average concentration of RM-718 during a dosing interval in steady state
t1/2 measurement of RM-718 | up to 168 hours post-dose on Day 1 (Parts A, B and C) and 168 hours post-dose on Day 22 (Parts B and C).
  Terminal elimination half-life of RM-718 in plasma
λz measurement of RM-718 | up to 168 hours post-dose on Day 1 (Parts A, B and C) and 168 hours post-dose on Day 22 (Parts B and C).
  Estimate of the terminal elimination rate constant of RM-718
CL/F measurement of RM-718 | up to 168 hours post-dose on Day 1 (Parts A, B and C) and 168 hours post-dose on Day 22 (Parts B and C).
  Clearance of RM-718 following extravascular administration
Vz/F measurement of RM-718 | up to 168 hours post-dose on Day 1 (Parts A, B and C) and 168 hours post-dose on Day 22 (Parts B and C).
  Volume of distribution of RM-718 following extravascular administration
Accumulation ratio of RM-718 | Week 1 to Week 4 (AUC on Week 4/AUC on Week 1) (Parts B, C)
  Ratio of accumulation of RM-718 under steady state conditions
Change from baseline in BMI (Part C only) | Baseline to Week 16
Mean change in weight (Part C only) | Baseline to Week 16
Mean change in waist circumference (Part C only) | Baseline to Week 16
Mean change in weekly average of the daily most hunger score in patients ≥12 years of age (Part C only) | Baseline to Week 16
Mean change in weekly average of the Symptoms of Hyperphagia composite score (Part C only) | Baseline to Week 16
Ctrough measurement of RM-718 (Part D) | up to 168 hours post-dose on Day 8 and up to 168 hours post-dose on Day 29
  Observed pre-dose plasma concentration of RM-718
Change from baseline in BMI (Part D) | Baseline to Week 26
Mean change in weight (Part D) | Baseline to Week 26
Mean change in waist circumference (Part D) | Baseline to Week 26
Mean change in the weekly average of the Prader-Willi Syndrome Food Problem Diary (PWS-FPD) total score (Part D) | Baseline to Week 26
Mean change in the Hyperphagia Questionnaire for Clinical Trials (HQ-CT) total score (Part D) | Baseline to Week 26
Change in total body mass (Part D) | Baseline to Week 26
  Change in body mass as measured by dual-energy x-ray

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (7):
- United States (7):
  - UAB Pediatric Endocrinology (Part C and Part D), Birmingham, Alabama
  - Ann and Robert H. Lurie Children's Hospital of Chicago (Part C and Part D), Chicago, Illinois
  - Boston Children's Hospital (Part C only), Boston, Massachusetts
  - Brigham and Women's Hospital (Part C and Part D), Boston, Massachusetts
  - Vanderbilt University Medical Center (Part C only), Nashville, Tennessee
  - Worldwide Clinical Trials (Part A and Part B), San Antonio, Texas
  - University of Utah Pediatric Endocrine Clinic (Part C and Part D), Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No